CLINICAL TRIAL: NCT02669446
Title: Non Interventional Clinical Investigation of Ectoin® Lozenges in the Treatment of Acute Viral Pharyngitis
Brief Title: Ectoin® Lozenges in the Treatment of Acute Viral Pharyngitis
Status: Completed | Type: Observational
Sponsor: Bitop AG (Industry)
Responsible Party: Sponsor
Other Study IDs: 2016/EHT/NIS
Record Dates: First submitted 2016-01-21; First posted 2016-02-01 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Acute Viral Pharyngitis
Keywords: Non interventional study; Ectoin; Lozenges; pharyngitis
MeSH Terms: conditions — Pharyngitis | interventions — Equipment and Supplies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Ectoin containing Lozenges: treatment with Ectoin containing lozenges
  Interventions: Device: Medical devices
- Hyaluronic acid containing lozenges: treatment with hyaluronic acid containing lozenges
  Interventions: Device: Medical devices
- Saline solution for gargling: Subjects in were requested to gargle with salt water
  Interventions: Device: traditional household remedy

INTERVENTIONS:
Device: Medical devices
  Groups: Ectoin containing Lozenges; Hyaluronic acid containing lozenges
Device: traditional household remedy
  Groups: Saline solution for gargling

SUMMARY:
This a comparative, open label, parallel group, non interventional study which compares the tolerability and influence of Ectoin containing Lozenges to saline solution and lozenges containing hyaluronic acid for the treatment of acute viral Pharyngitis. The observation takes place over a period of 7 days. Response to treatment is recorded at day 1 and day 7 by the physician and by the patient in a dairy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute Pharyngitis according to instruction for use
* Female or male individuals ≥ 18 years
* Agreement to abide by the routinely provided doctor's appointment for follow- up (reflected in the planned visits of observation plan resist)

Exclusion Criteria:

* Contraindications according to instructions for use
* Male or female person under 18 years
* Sore throat for more than 5 days
* Any disease that can, in the opinion of the treating physician to affect the outcome of the study.
* Patients with known intolerance to one of the substances used
* Surgical procedures to the mouth and throat in the last 6 weeks before inclusion in the NIS
* Bacterial Pharyngitis
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with viral pharyngitis
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2016-01; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in Pharyngitis symptom score evaluated by the physician | day 1 and day 7
  The intensity of the symptoms and signs will be graded on a continuous numeric scale, i.e. absent-0, severe-10.
  The following signs and symptoms will be documented:
  * pain on swallowing
  * tickle in the throat
  * hoarseness
  * dry mouth and throat
  * burning of throat
  * patient´s General condition
  * reddening of the oropharynx
  * reddening of the larynx

SECONDARY OUTCOMES:
Change in Pharyngitis symptoms evaluated on patient´s diaries | 7 days
  The intensity of the symptoms and signs will be graded on a continuous numeric scale, i.e. absent-0, severe-10.
  The following signs and symptoms will be documented:
  * pain on swallowing
  * tickle in the throat
  * hoarseness
  * dry mouth and throat
  * burning of throat
  * patient´s General condition
Change in patient´s General condition evaluated by the physician | day 1 and day 7
Patient´s Evaluation of tolerability | 7 days
  Assessment of tolerability on a numeric scale (bad-0; very good-10)
physician´s Evaluation of tolerability | day 7
  Assessment of tolerability on a numeric scale (bad-0; very good-10)
Change in number and type of adverse Events | 7 days
  Incidence of adverse Events and correlations with the therapy

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Sonnemann, MD, Principal Investigator — HNO-Praxis
Locations (4):
- Germany (4):
  - HNO-Praxis Elmshorn, Elmshorn, Elmshorn
  - HNO-Praxis Mahlstedt, Berlin
  - HNO-Praxis Möller, Lüneburg
  - HNO-Praxis, Norderstedt